CLINICAL TRIAL: NCT05626010
Title: Efficacy of Acetaminophen-ibuprofen Combination on the Postoperative Pain After Thyroidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Young Eun Moon, professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAP-ibuprofen-thyroid
Record Dates: First submitted 2022-11-15; First posted 2022-11-23 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Thyroid Disease
MeSH Terms: conditions — Thyroid Diseases | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): acetaminophen 1g iv dripping
  Interventions: Drug: Acetaminophen
- experimental group (Experimental): the combination of acetaminophen 1g and ibuprofen 300mg iv dripping
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen

INTERVENTIONS:
Drug: Acetaminophen — acetaminophen 1g iv dripping at end of surgery
Drug: Ibuprofen — ibuprofen 300mg iv dripping at end of surgery
  Arms: experimental group

SUMMARY:
Acetaminophen and ibuprofen has been safely used for a long time and reduces postoperative pain and opioid dosages. Investigators are planning to compare the efficacy of 1) acetaminophen only and 2) acetaminophen and ibuprofen combination at postoperative pain after thyroidectomy.

DETAILED DESCRIPTION:
Acetaminophen and ibuprofen has been safely used for a long time and reduces postoperative pain and opioid dosages. Investigators are planning to compare the efficacy of 1) acetaminophen 1g only and 2) the combination of acetaminophen 1g and ibuprofen 300mg at postoperative pain after thyroidectomy. Some recovery valuables such as the postoperative pain and opioid requirements will be assessed

ELIGIBILITY:
Inclusion Criteria:

* the patients undergoing scheduled thyroidectomy
* American Society of Anesthesiologists status 1 or 2

Exclusion Criteria:

* refusal to be enrolled in the study
* emergency surgery
* hepatic or renal disease
* on chronic pain medications
* psychiatric disorders
* pregnancy, lactation
* allergy or contraindication to the study drug

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | during 30 minutes after surgery
  the maximal postoperative pain severity using pain scale(visual analogue scale; 0 cm=no pain; 10 cm=the worst pain)

SECONDARY OUTCOMES:
pain killer requirement | during 30 minutes after surgery
  the incidence of the patients who require pain killer

CONTACTS AND LOCATIONS:
Overall Officials: youngeun moon, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, Seocho-gu, South Korea

IPD SHARING:
Plan to Share IPD: No